CLINICAL TRIAL: NCT03880227
Title: Improving Visual Attention to Social Stimuli in Individuals With Schizophrenia
Brief Title: Improving Visual Attention in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, Hans Klein, Principal Investigator, The University of Texas at Dallas
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 19-58
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Results first posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be paired based on key demographic criteria and assigned to one of two stimulation locations (rTPJ or dmPFC), participants will then complete active and sham stimulation sessions in a randomized, counterbalanced order approximately one week apart.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Anodal followed by sham stimulation tDCS to rTPJ (Experimental): cross-over design - active stimulation tDCS to the rTPJ followed by behavioral testing. After 1 week washout, sham stimulation tDCS to the rTPJ followed by behavioral testing.
  Interventions: Device: Active anodal tDCS; Device: Sham tDCS
- Anodal followed by sham stimulation tDCS to dmPFC (Active Comparator): cross-over design - active stimulation tDCS to the dmPFC followed by behavioral testing. After 1 week washout, sham stimulation tDCS to the dmPFC followed by behavioral testing.
  Interventions: Device: Active anodal tDCS; Device: Sham tDCS
- Sham followed by anodal stimulation tDCS to rTPJ (Experimental): cross-over design - sham stimulation tDCS to the rTPJ followed by behavioral testing. After 1 week delay, active stimulation tDCS to the rTPJ followed by behavioral testing.
  Interventions: Device: Active anodal tDCS; Device: Sham tDCS
- Sham followed by anodal stimulation tDCS to dmPFC (Active Comparator): cross-over design - sham stimulation tDCS to the dmPFC followed by behavioral testing. After 1 week delay, active stimulation tDCS to the dmPFC followed by behavioral testing.
  Interventions: Device: Active anodal tDCS; Device: Sham tDCS

INTERVENTIONS:
Device: Active anodal tDCS — active anodal tDCS with behavioral tasks to assess visual attention
Device: Sham tDCS — sham tDCS with behavioral tasks to assess visual attention

SUMMARY:
This study investigates whether visual attention can be improved in individuals with schizophrenia by stimulating the brain via transcranial Direct Current Stimulation (tDCS).

DETAILED DESCRIPTION:
Individuals with schizophrenia tend to display abnormal visual attention when performing visual tasks, typically spending less time on salient features of the stimuli (e.g. core facial features or body movement in social tasks), and instead focusing on idiosyncratic features of an image or video. Poor visual attention in schizophrenia has been directly linked to poorer social cognitive performance (e.g. recognizing emotional expressions or social cues) which can impact an individual's day to day functioning.

Transcranial Direct Current Stimulation (tDCS) is a form of noninvasive neurostimulation which has been proposed as a therapeutic procedure in numerous psychiatric disorders. TDCS in schizophrenia has been demonstrated to improve a wide range of cognitive processes, and in healthy adults, tDCS has been demonstrated to improve aspects of social cognition. TDCS thus appears to be a promising therapeutic technique that may be useful for improving visual attention in patients with schizophrenia, and potentially impact social cognitive performance via an underlying mechanism tying the two. This study will compare visual performance in individuals with schizophrenia across two conditions: active anodal tDCS and sham tDCS, while also comparing between brain stimulation sites: rTPJ and dmPFC.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV-TR or DSM-5 diagnosis of schizophrenia or schizoaffective disorder and clinically stable (i.e. no hospitalizations) for at least 8 weeks prior to informed consent and be on a stable medication regimen for at least 6 weeks with no dose changes for a minimum of 2 weeks prior to informed consent.

Exclusion Criteria:

* The presence or history of a pervasive developmental disorder or mental retardation as defined by a premorbid IQ < 70
* Presence or history of medical or neurological disorders in which neural stimulation would be contraindicated (e.g. presence of epilepsy or history of seizures)
* Presence of sensory limitations, including visual or hearing impairments that interfere with assessment
* History of electroconvulsive therapy
* Not proficient in English
* Presence of substance abuse in the past one month or dependence not in remission in the past six months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans S Klein, MS, Principal Investigator — The University of Texas at Dallas
Locations (1):
- The University of Texas at Dallas, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 81 participants were recruited to the study between March 2019 and March 2020 at a university site in Dallas, TX.
Pre-assignment Details: At enrollment, all participants were matched in pairs based upon key demographic factors (i.e., age, race, gender, and education), and pairs were randomly assigned to stimulation condition, resulting in separate rTPJ and dmPFC stimulation groups. 5 participants did not complete both study visits, with 4 participants not returning to their second visit, and 1 participant discontinuing their first visit prior to stimulation procedures.
Groups:
- Anodal Followed by Sham Stimulation tDCS to rTPJ: Active stimulation tDCS over the rTPJ followed by behavioral testing. Active Stimulation: 2mA for 20 minutes (15s ramp up and ramp down)
  After 1 week washout, sham stimulation tDCS to the rTPJ followed by behavioral testing Sham stimulation: pre-programmed sham condition, direct current for 30 seconds, intermittent impedance control checks during the remainder of the 20-minutes
- Anodal Followed by Sham Stimulation tDCS to dmPFC: Active stimulation tDCS over the dmPFC followed by behavioral testing. Active Stimulation: 2mA for 20 minutes (15s ramp up and ramp down)
  After 1 week washout, sham stimulation tDCS to the dmPFC followed by behavioral testing Sham stimulation: pre-programmed sham condition, direct current for 30 seconds, intermittent impedance control checks during the remainder of the 20-minutes
- Sham Followed by Anodal Stimulation tDCS to rTPJ: Sham stimulation tDCS to the rTPJ followed by behavioral testing Sham stimulation: pre-programmed sham condition, direct current for 30 seconds, intermittent impedance control checks during the remainder of the 20-minutes
  After 1 week delay, Active stimulation tDCS over the rTPJ followed by behavioral testing.
  Active Stimulation: 2mA for 20 minutes (15s ramp up and ramp down)
- Sham Followed by Anodal Stimulation tDCS to dmPFC: Sham stimulation tDCS to the dmPFC followed by behavioral testing Sham stimulation: pre-programmed sham condition, direct current for 30 seconds, intermittent impedance control checks during the remainder of the 20-minutes
  After 1 week delay, Active stimulation tDCS over the dmPFC followed by behavioral testing.
  Active Stimulation: 2mA for 20 minutes (15s ramp up and ramp down)
Period: First Visit
Arm/Group | Anodal Followed by Sham Stimulation tDCS to rTPJ | Anodal Followed by Sham Stimulation tDCS to dmPFC | Sham Followed by Anodal Stimulation tDCS to rTPJ | Sham Followed by Anodal Stimulation tDCS to dmPFC
Started | 20 | 21 | 22 | 18
Completed | 19 | 21 | 22 | 18
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: 1 Week Washout/ Delay
Arm/Group | Anodal Followed by Sham Stimulation tDCS to rTPJ | Anodal Followed by Sham Stimulation tDCS to dmPFC | Sham Followed by Anodal Stimulation tDCS to rTPJ | Sham Followed by Anodal Stimulation tDCS to dmPFC
Started | 19 | 21 | 22 | 18
Completed | 19 | 20 | 19 | 18
Not Completed | 0 | 1 | 3 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0
Not completed — Incompatibility with technical component (eyetracking) | 0 | 0 | 1 | 0
Period: Second Visit
Arm/Group | Anodal Followed by Sham Stimulation tDCS to rTPJ | Anodal Followed by Sham Stimulation tDCS to dmPFC | Sham Followed by Anodal Stimulation tDCS to rTPJ | Sham Followed by Anodal Stimulation tDCS to dmPFC
Started | 19 | 20 | 19 | 18
Completed | 19 | 20 | 19 | 18
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Anodal/Sham Stimulation tDCS to rTPJ: Within subject design - sham and anodal tDCS to the rTPJ followed by behavioral testing
  Active anodal tDCS: active anodal tDCS with behavioral tasks to assess visual attention Sham tDCS: sham tDCS with behavioral tasks to assess visual attention
- Anodal/Sham Stimulation tDCS to dmPFC: Within subject design - sham and anodal tDCS to the dmPFC followed by behavioral testing
  Active anodal tDCS: active anodal tDCS with behavioral tasks to assess visual attention Sham tDCS: sham tDCS with behavioral tasks to assess visual attention
- Total: Total of all reporting groups
Arm/Group | Anodal/Sham Stimulation tDCS to rTPJ | Anodal/Sham Stimulation tDCS to dmPFC | Total
Number analyzed (Participants) | 42 | 39 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 39 | 81
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.74 (10.58) | 40.79 (11.55) | 40.77 (10.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 23 | 21 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 35 | 33 | 68
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 22 | 47
  White | 17 | 14 | 31
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 39 | 81

OUTCOME MEASURES:

1. Primary Outcome: Visual Attention to Static Faces
Description: Visual attention measured via eye-tracking (percentage of time attending to investigator designated AOIs) when viewing static, emotional faces (stimuli: Emotion Recognition - 40). AOIs for static faces will be defined as core facial features (i.e. eyes, nose, mouth).
Time Frame: Assessment will be completed 30 minutes after completion of the active/sham stimulation
Population: Population analyzed were those that completed both active and sham stimulations (n=5 removed) with valid eyetracking data (n=2 removed)
Measure: Mean (Standard Deviation); unit: proportion of time attending to AOIs
Groups:
- Anodal Stimulation tDCS to rTPJ: anodal tDCS to the rTPJ followed by behavioral testing
  Active anodal tDCS: active anodal tDCS with behavioral tasks to assess visual attention
- Sham tDCS to rTPJ: sham tDCS to the rTPJ followed by behavioral testing
  Sham tDCS: sham tDCS with behavioral tasks to assess visual attention
- Anodal Stimulation tDCS to dmPFC: anodal tDCS to the dmPFC followed by behavioral testing
  Active anodal tDCS: active anodal tDCS with behavioral tasks to assess visual attention
- Sham tDCS to dmPFC: sham tDCS to the dmPFC followed by behavioral testing
  Sham tDCS: sham tDCS with behavioral tasks to assess visual attention
Arm/Group | Anodal Stimulation tDCS to rTPJ | Sham tDCS to rTPJ | Anodal Stimulation tDCS to dmPFC | Sham tDCS to dmPFC
Number analyzed (Participants) | 37 | 37 | 37 | 37
proportion of time attending to AOIs | 0.54 (0.15) | 0.52 (0.15) | 0.57 (0.13) | 0.53 (0.14)

2. Primary Outcome: Visual Attention to Dynamic Actor
Description: Visual attention measured via eye-tracking(percentage of time attending to investigator designated AOIs) when viewing videos of a single actor (stimuli: Bell Lysaker Emotion Recognition Task). AOIs for this task will be defined as core facial features (i.e. eyes, nose, and mouth).
Time Frame: Assessment will be completed 30 minutes after completion of the active/sham stimulation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: proportion of time attending to AOIs
Arm/Group | Anodal Stimulation tDCS to rTPJ | Sham tDCS to rTPJ | Anodal Stimulation tDCS to dmPFC | Sham tDCS to dmPFC
Number analyzed (Participants) | 37 | 37 | 37 | 37
proportion of time attending to AOIs | 0.47 (0.12) | 0.46 (0.11) | 0.47 (0.11) | 0.47 (0.11)

3. Primary Outcome: Visual Attention to Dynamic Social Scenes
Description: Visual attention measured via eye-tracking (percentage of time attending to investigator designated AOIs) when viewing videos of two or more actors in a scene (stimuli: The Awareness of Social Inference Task Part 3, Version A). AOIs for this task will be defined as salient social and contextual stimuli (e.g. social stimuli are faces of actors, while contextually salient stimuli include items actors are talking about, such as a plate full of food or an empty wallet).
Time Frame: Assessment will be completed 30 minutes after completion of the active/sham stimulation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: proportion of time attending to AOIs
Arm/Group | Anodal Stimulation tDCS to rTPJ | Sham tDCS to rTPJ | Anodal Stimulation tDCS to dmPFC | Sham tDCS to dmPFC
Number analyzed (Participants) | 37 | 37 | 37 | 37
proportion of time attending to AOIs | 0.22 (0.06) | 0.23 (0.07) | 0.26 (0.07) | 0.25 (0.07)

4. Secondary Outcome: Fixation Stabilization
Description: Stabilization of visual fixation on fixation circle positioned in middle of screen. Participants will be placed in front of an eyetracking device and asked to keep their eyes focused on a circle in the middle of the screen. Stabilization will be measured via eye-tracking as the deviation from a single point on screen, calculated by assessing the sum of squares of both the x and y axis (output from eyetracking device). Higher number indicates more movement, and thus less stabilization.
Time Frame: Assessment will be completed 30 minutes after completion of the active/sham stimulation
Population: Population analyzed were those that completed both active and sham stimulations (n=6 removed) with valid eyetracking data (n=2 removed)
Measure: Mean (Standard Deviation); unit: pixels (equivalent: 1/96th in or 0.26mm)
Arm/Group | Anodal Stimulation tDCS to rTPJ | Sham tDCS to rTPJ | Anodal Stimulation tDCS to dmPFC | Sham tDCS to dmPFC
Number analyzed (Participants) | 37 | 37 | 36 | 36
pixels (equivalent: 1/96th in or 0.26mm) | 0.10 (0.24) | 0.08 (0.14) | 0.05 (0.10) | 0.07 (0.14)

ADVERSE EVENTS:
Time Frame: From time of visit 1 through the follow up phone call (Average time around 10 days, longest duration 29 days)
Description: Routine effects of tDCS were assessed during visit and in follow up phone calls performed after scheduled visits. Definition of adverse events are any events that were beyond these typically reported events.
Arm/Group | Anodal Stimulation tDCS to rTPJ | Sham tDCS to rTPJ | Anodal Stimulation tDCS to dmPFC | Sham tDCS to dmPFC
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/41 | 0/39 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/41 | 0/39 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 1/41 | 0/39 | 0/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anodal Stimulation tDCS to rTPJ (N=38) | Sham tDCS to rTPJ (N=41) | Anodal Stimulation tDCS to dmPFC (N=39) | Sham tDCS to dmPFC (N=38)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — participant voluntarily reported experiencing a migraine a few days after sham tDCS visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT03880227/Prot_SAP_001.pdf